CLINICAL TRIAL: NCT07021612
Title: A Clinical and Imaging Registry of Transcatheter Aortic Valve Implantation Using JenaValve System/ J-Valve System for Patients With Pure Aortic Regurgitation: An Observational Study
Brief Title: A Clinical and Imaging Registry of Transcatheter Aortic Valve Implantation Using JenaValve System/ J-Valve System for Patients With Pure Aortic Regurgitation
Acronym: CAIR-JAR
Status: Recruiting | Type: Observational
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr So Chak Yu kent, Clinical Assistant Professor, Prince of Wales Hospital, Shatin, Hong Kong
Other Study IDs: 2025.079
Record Dates: First submitted 2025-06-05; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Aortic Valve Disease
Keywords: Transcatherter Aortic Valve Intervention
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Interventional group: Patient implanted with J-Valve or JenaValve TAVI system
  Interventions: Device: JenaValve; Device: J-Valve

INTERVENTIONS:
Device: JenaValve — JenaValve is a newly developed advanced TAVI system developed by Jenavalve Technology Inc.
Device: J-Valve — J-Valve is a newly developed advanced TAVI system developed by Genesis Medtech.

SUMMARY:
Aortic regurgitation (AR) is not uncommon. Transcatheter aortic valve implantation (TAVI) for treating pure aortic regurgitation is a potential future treatment option for pure AR especially in patients having high risk for open heart surgery.

TAVI using dedicated device for pure AR has a different anchor mechanism to TAVI for aortic stenosis (AS). AR patientsalso have different cardiac flow pattern, aortic root pathology and left ventricular remodeling pattern compared to AS patients. Subclinical leaflet thrombosis has been described in AS patient receiving TAVI, which will affect the durability and antithrombotic regime. Follow-up imaging for dedicated TAVI device in AR patient is limited.

ELIGIBILITY:
Inclusion Criteria:

1. receiving transcatheter aortic valve implantation (TAVI) (using Jenavalve/J-Valve) in PWH
2. with severe symptomatic AR (NYHA III-IV) despite optimal medical therapy
3. Deemed high risk for aortic valve surgery determined by a multidisciplinary heart team (including cardiologists, cardiac surgeons and cardiac anesthetists)
4. Capable of providing informed consent

Exclusion Criteria:

1. Evidence of intracardiac mass, thrombus or vegetation
2. Anatomical structures precluding proper device deployment or device vascular access, evaluated by echo or CT
3. Sepsis or active endocarditis within 3 months, or infections requiring antibiotic therapy within 2 weeks prior to the planned procedure
4. Subjects currently participating in another clinical trial of an investigational drug or device that has not yet completed its primary endpoint.
5. Chronic Kidney Disease with eGFR <30 ml/min/1.73m2.
6. Cardiogenic shock or other hemodynamic instability requiring inotropic support or ventricular assist device
7. Contraindicated for CT or MRI assessment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients receiving transcatheter aortic valve implantation (TAVI) (using Jenavalve/J-Valve) in PWH with severe symptomatic AR (NYHA III-IV) despite optimal medical therapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Presence of leaflet thrombosis | 6 month
  Presence of hypoattenuated leaflet thickening (HALT) detected on 6 month follow-up computed tomography
Presence of leaflet thrombosis | 6 month
  Presence of restricted leaflet motion (RELM) detected on 6 month follow-up computed tomography
Presence of leaflet thrombosis | 6 month
  Presence of hypoattenuation affecting motion (HAM) detected on 6 month follow-up computed tomography

SECONDARY OUTCOMES:
Magnetic Resonance Imaging (MRI) | 1 month
  Comparison of 4D-Flow pattern using MRI at 1 month post-OP vs pre-OP
Magnetic Resonance Imaging (MRI) | 1 month
  Comparison of Aortic Valve Flow Velocity using MRI at 1 month post-OP vs pre-OP
Magnetic Resonance Imaging (MRI) | 1 month
  Comparison of Aortic Wall shear stress using MRI at 1 month post-OP vs pre-OP
Magnetic Resonance Imaging (MRI) | 1 month
  Comparison of Intraventricular flow pattern using MRI at 1 month post-OP vs pre-OP
Computed Tomographic Endpoints | Baseline
  Presence of leaflet thrombosis (hypoattenuated leaflet thickening (HALT) on CT images at baseline
Computed Tomographic Endpoints | Up to 1-month post-OP
  Presence of leaflet thrombosis (hypoattenuated leaflet thickening (HALT) on CT images at post-OP
Computed Tomographic Endpoints | 1-year
  Presence of leaflet thrombosis (hypoattenuated leaflet thickening (HALT) on CT images at 1 year post-OP
Computed Tomographic Endpoints | Baseline
  Presence of leaflet thrombosis (restricted leaflet motion (RELM)) on CT images at baseline
Computed Tomographic Endpoints | Up to 1-month post-OP
  Presence of leaflet thrombosis (restricted leaflet motion (RELM)) on CT images at post-OP
Computed Tomographic Endpoints | 1-year
  Presence of leaflet thrombosis (restricted leaflet motion (RELM)) on CT images at 1 year post-OP
Computed Tomographic Endpoints | Baseline
  Presence of leaflet thrombosis (hypoattenuation affecting motion (HAM )on CT images at baseline
Computed Tomographic Endpoints | Upto 1-month post-OP
  Presence of leaflet thrombosis (hypoattenuation affecting motion (HAM )on CT images at post-OP
Computed Tomographic Endpoints | 1-year
  Presence of leaflet thrombosis (hypoattenuation affecting motion (HAM )on CT images at 1 year post-OP
Computed Tomographic Endpoints | Baseline
  To obtain the native valve dimensions using CT imaging at pre-OP (baseline)
Computed Tomographic Endpoints | Up to 1-month post-OP
  To compare the impanted Transcatheter valve dimensions using CT imaging with baseline at post-OP
Computed Tomographic Endpoints | 6-month
  To compare the impanted Transcatheter valve dimensions using CT imaging with baseline at 6 month post-OP
Computed Tomographic Endpoints | 1-year
  To compare the impanted Transcatheter valve dimensions using CT imaging with baseline at 12 month post-OP
Computed Tomographic Endpoints | Up to 1-month post-OP
  To obtain the impanted Transcatheter valve location using CT imaging at post-OP
Computed Tomographic Endpoints | 6-month
  To compare the impanted Transcatheter valve location using CT imaging with post-OP at 6 month post-OP
Computed Tomographic Endpoints | 1-year
  To compare the impanted Transcatheter valve location using CT imaging with post-OP at 12 month post-OP
Computed Tomographic Endpoints | Baseline
  To obtain the native valve leaflet overhang using CT imaging at pre-OP (baseline)
Computed Tomographic Endpoints | Up to 1-month post-OP
  To obtain the impanted valve leaflet overhang using CT imaging at post-OP
Computed Tomographic Endpoints | 6-month
  To compare the impanted valve leaflet overhang using CT imaging with post-OP at 6 month post-OP
Computed Tomographic Endpoints | 1-year
  To compare the impanted valve leaflet overhang using CT imaging with post-OP at 12 month post-OP
Echocardiographic Endpoints | Baseline
  To grade AR Severity using echocardiography at baseline ii. Mean Aortic valve pressure gradient iii. Left Ventricular Ejection Fraction (LVEF) iv. Paravalvular leak severity
Echocardiographic Endpoints | day 1-7
  To grade AR Severity using echocardiography at Day 1-7 post-OP
Echocardiographic Endpoints | day 30
  To grade AR Severity using echocardiography at Day30 post-OP
Echocardiographic Endpoints | 6-month
  To grade AR Severity using echocardiography at 6 months post-OP
Echocardiographic Endpoints | 1-year
  To grade AR Severity using echocardiography at 1 year post-OP
Echocardiographic Endpoints | Baseline
  To obtain Mean Aortic valve pressure gradient using echocardiography at baseline
Echocardiographic Endpoints | day 1-7
  To obtain Mean Aortic valve pressure gradient using echocardiography at Day 1-7 post OP
Echocardiographic Endpoints | day 30
  To obtain Mean Aortic valve pressure gradient using echocardiography at Day 30 post OP
Echocardiographic Endpoints | 6-month
  To obtain Mean Aortic valve pressure gradient using echocardiography at 6 months post OP
Echocardiographic Endpoints | 1-year
  To obtain Mean Aortic valve pressure gradient using echocardiography at 12 months post OP
Echocardiographic Endpoints | Baseline
  To obtain Left Ventricular Ejection Fraction (LVEF) using echocardiography at baseline
Echocardiographic Endpoints | Day 1-7 post OP
  To obtain Left Ventricular Ejection Fraction (LVEF) using echocardiography at Day 1-7 post OP
Echocardiographic Endpoints | Day30 post OP
  To obtain Left Ventricular Ejection Fraction (LVEF) using echocardiography at Day 30 post OP
Echocardiographic Endpoints | 6 months post OP
  To obtain Left Ventricular Ejection Fraction (LVEF) using echocardiography at 6 months post OP
Echocardiographic Endpoints | 12 months post OP
  To obtain Left Ventricular Ejection Fraction (LVEF) using echocardiography at 12 months post OP
Echocardiographic Endpoints | Day 1-7 post OP
  To evaluate Paravalvular leak severity using echocardiography at Day 1-7 post OP
Echocardiographic Endpoints | Day 30 post OP
  To evaluate Paravalvular leak severity using echocardiography at Day 30 post OP
Echocardiographic Endpoints | 6 months post OP
  To evaluate Paravalvular leak severity using echocardiography at 6 months post OP
Echocardiographic Endpoints | 12 months post OP
  To evaluate Paravalvular leak severity using echocardiography at 12 months post OP
cardiovascular Mortality events | 12 months post OP
  cardiovascular Mortality event up till 12 months post-OP
Myocardial Infarction event | 12 months post OP
  Myocardial Infarction (MI) event up till 12 months post-OP
Stroke event | 12 months post OP
  Stroke event up till 12 months post-OP
New onset renal failure event | 12 months post OP
  New onset renal failure requiring unplanned dialysis or renal replacement therapyevent up till 12 months post-OP
Severe Bleeding event | 12 months post OP
  Severe Bleeding (includes fatal, life-threatening and extensive bleeding as defined by VARC) event up till 12 months post-OP
Non-elective aortic valve surgery event | 12 months post OP
  Non-elective aortic valve surgery event up till 12 months post-OP
Non-elective transcatheter re-intervention event | 12 months post OP
  Non-elective transcatheter re-intervention post procedure event up till 12 months post-OP
Major cardiac structural complications | 12 months post OP
  Major cardiac structural complications event up till 12 months post-OP
Major access site complications | 12 months post OP
  Major access site complications event up till 12 months post-OP
New pacemaker implantation event | 12 months post OP
  New pacemaker implantation due to AV block event up till 12 months post-OP
Acute Device Success Rate | immediately post-OP
  Rate of successful deployment of the device and removal of the delivery system as planned, with no unplanned surgery related to the device or access procedure immediately post-OP
Procedural Success Rate | immediately post-OP
  Rate of Device success without clinically significant PVL, as determined by the Echo Core Lab (ECL) assessment of a discharge TTE. Subjects who die or undergo aortic valve surgery before discharge are procedure failures.
All-cause mortality | 30-day
  30-day all-cause mortality rate of subjects
All-cause mortality | 1-year
  1-year all-cause mortality rate of subjects
heart failure hospitalization | 30-day
  30-day heart failure hospitalization rate of subjects
heart failure hospitalization | 1-year
  1 year heart failure hospitalization rate of subjects
NYHA Functional Class | Baseline
  NYHA Functional Class of subjects at baseline
NYHA Functional Class | Post-OP
  NYHA Functional Class of subjects at post-OP
NYHA Functional Class | 1 month Post-OP
  NYHA Functional Class of subjects at 1 month post-OP
NYHA Functional Class | 6-month Post-OP
  NYHA Functional Class of subjects at 6-month post-OP
NYHA Functional Class | 12-month Post-OP
  NYHA Functional Class of subjects at 12-month post-OP

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong